CLINICAL TRIAL: NCT03307434
Title: PREVATHLE: To Evaluate the Effectiveness of an Injury Prevention Program in Athletics
Brief Title: To Evaluate the Effectiveness of an Injury Prevention Program in Athletics
Acronym: PREVATHLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1708116; ID-RCB (Other: 2017-A01980-53)
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-09

CONDITIONS: Athletics; Wounds and Injuries; Prevention Program
Keywords: Program; Prevention; Injury; Athletics
MeSH Terms: conditions — Wounds and Injuries | interventions — 2-amino-5-iodo-6-phenyl-4-pyrimidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): experimental group is composed of athletes will be followed the Athletics Injury Prevention Program
  Interventions: Other: Athletics Injury Prevention Program
- control group (Active Comparator): control group is composed of athletes will be continued their regular training
  Interventions: Other: regular training

INTERVENTIONS:
Other: Athletics Injury Prevention Program — The Athletics Injury Prevention Program (AIPP) will be performed by experimental group twice a week. The AIPP is composed of 8 exercises including core stability, balance, pelvic stabilization, stretching and strengthening of the Achilles tendon and hamstrings.
  Other Names: AIPP
  Arms: experimental group
Other: regular training — The regular training will be performed by control group according to the standard practice.
  Other Names: standard practice
  Arms: control group

SUMMARY:
The practice of Athletics leads to risk of injuries: about 61 to 76% athletes will occurred at least one injury during a season. The prevention of Athletics injuries thus represents a major challenge for all stakeholders around athletes. In team sports, injury prevention programs have been implemented and scientifically validated. However, no injury prevention programs have been implemented and scientifically validated for Athletics. In this context, a primary objective will be to analyze the effectiveness of an Athletics Injury Prevention Program (AIPP) to reduce the frequency (percentage) of athletes presenting at least one injury complaint related to athletic practice at long term (40 weeks). A statistician will carry out a randomized control trial in cluster (clubs with AIPP and clubs without AIPP), multicenter, including athletes between 15 and 40 years old and licensed in athletic clubs and followed during an athletic season.

DETAILED DESCRIPTION:
The person in charge of the platform will collect on a weekly basis via a IT-questionnaire sent out automatically every Monday the following parameters: injury complaints (presence or absence, and characteristics if presence) and exposure (number of hours of athletic practice (training and competition) and intensity), and the number of AIPP realization per week. The main criterion will be the frequency (percentage) of athletes presenting at least one injury complaint that have a consequence on the practice (reduction or cessation of practice).

ELIGIBILITY:
Inclusion Criteria:

* To dismissed in athletics clubs affiliated to French Federation of Athletics
* To practice one of the disciplines of athletics
* Men or women aged between 15 and 40 years

Exclusion Criteria:

- Patient's refusal to participate in the study and / or inability to express agreement or signing the informed consent

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 880 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
injury complaint and have a consequence on the practice | at 40 weeks
  Frequency of athletes presenting at least one injury complaint and have a consequence on the practice (reduction or cessation of practice).

SECONDARY OUTCOMES:
injury complaint number and hours number of athletic practice | at 40 weeks
  Correlation between injury complaint number and hours number of athletic practice
injury complaint number and weeks number of athletic practice | at 40 weeks
  Correlation between injury complaint number and weeks number of athletic practice
week without injury complaints | at 40 weeks
  Frequency of week without injury complaints
injury complaint number at the training | at 40 weeks
  Frequency of injury complaint number at the training
injury complaint number and at the competition | at 40 weeks
  Frequency of injury complaint number at the competition
type of injury complaint between 4 consequences | at 40 weeks
  the 4 consequences of injury complaint are : No consequence of athletic practice; reduce practice; Stop practice; and Consequence of practice
injury complaint number by groups | at 40 weeks
  Correlation of injury complaint number by groups
injury complaint type | at 40 weeks
  Number of injury complaint type: hamstrings, Achilles tendons, ankles, knees and rachis

CONTACTS AND LOCATIONS:
Overall Officials: Pascal EDOUARD, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iatropoulos S, Dandrieux PE, Navarro L, Blanco D, Edouard P. The Dose-Response Relationship of an Exercise-Based Injury Prevention Program: A Secondary Analysis of a Randomized Controlled Trial on Athletics (Track-and-Field) Athletes Over a 39-Week Follow-Up. Scand J Med Sci Sports. 2024 Sep;34(9):e14720. doi: 10.1111/sms.14720. PMID 39232249
- [Derived] Edouard P, Tondut J, Hollander K, Dandrieux PE, Navarro L, Bruneau A, Junge A, Blanco D. Risk factors for injury complaints leading to restricted participation in Athletics (Track and Field): a secondary analysis of data from 320 athletes over one season. BMJ Open Sport Exerc Med. 2023 Dec 7;9(4):e001718. doi: 10.1136/bmjsem-2023-001718. eCollection 2023. PMID 38089679
- [Derived] Edouard P, Steffen K, Peuriere M, Gardet P, Navarro L, Blanco D. Effect of an Unsupervised Exercises-Based Athletics Injury Prevention Programme on Injury Complaints Leading to Participation Restriction in Athletics: A Cluster-Randomised Controlled Trial. Int J Environ Res Public Health. 2021 Oct 28;18(21):11334. doi: 10.3390/ijerph182111334. PMID 34769849